CLINICAL TRIAL: NCT04914195
Title: Efficacy, Safety, and Pharmaco-kinetics of Leuprolide Acetate for Injection 3.75mg (Depot) (Leuprorelin) Administered in Subjects With Advanced Adenocarcinoma of Prostate: A Randomized, Active Controlled, Comparative, Open-Label, Multi-Center, Phase 3 Study
Brief Title: Leuprolide Acetate 3.75 mg Depot Injection for Patients With Advanced Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bharat Serums and Vaccines Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: BSV_LEUPR_18_05
Record Dates: First submitted 2021-05-31; First posted 2021-06-04 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Advanced Prostate Adenocarcinoma
MeSH Terms: interventions — Leuprolide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leuprolide acetate 3.75 mg Depot (Luprodex) (Experimental): Will be administered subcutaneously once a month for two cycles, on day 0 and on day 28/29
  Interventions: Drug: Leuprolide Acetate 3.75 MG/ML
- Leuprolide acetate 3.75 mg Depot (Lucrin) (Active Comparator): Will be administered subcutaneously once a month for two cycles, on day 0 and on day 28/29
  Interventions: Drug: Leuprolide Acetate 3.75 MG/ML

INTERVENTIONS:
Drug: Leuprolide Acetate 3.75 MG/ML — Leuprolide Acetate/ Leuprorelin is a depot injection administered as a subcutaneous injection once every month.

SUMMARY:
This is a Randomized, Active Controlled, Comparative, Open-Label, Multi-Center, Phase 3 clinical study to compare the efficacy, safety, and pharmacokinetics of leuprolide acetate for injection 3.75mg (depot) of two brands (Luprodex and Lucrin) administered in subjects with advanced adenocarcinoma of the prostate.

Approximately 168 subjects (males )of age above 18 years fulfilling the eligibility criteria will be enrolled. The IP will be given as a monthly dose for two cycles on day 0 and day 28.

The pharmacokinetic analysis will be done for 12 patients receiving Luprodex. The primary and secondary outcomes will be captured on days as per protocol. Adverse events will be noted for safety evaluation.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects aged above 18 years.
2. Histologically or cytologically confirmed adenocarcinoma of the prostate at stage T1b-4, Nany, Many in subjects, who would benefit from a GnRH agonist.
3. Baseline Testosterone of >1.50 ng/mL or >150 ng/dL.
4. For subjects with radical prostatectomy, an increase of 0.2 ng/mL or 20 ng/dL in PSA from previous test on two consecutive tests. For subjects with prostate irradiation a rise of greater than or equal to 2.0 ng/mL or 200 ng/dL PSA above the nadir.
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 (Appendix 2).
6. Life expectancy of at least 6 months from screening.
7. Adequate organ and immune system function
8. Willing to participate and sign the informed consent as per regulatory requirements.

Exclusion Criteria:

1. Evidence of brain metastases.
2. Evidence of spinal cord compression.
3. Evidence of urinary tract obstruction, where a flare in disease could put subject at significant risk in the opinion of the Investigator.
4. Received prostate cancer therapies like immunotherapy (antibody therapies, tumor vaccines), external radiotherapy, brachytherapy, chemotherapy or biological response modifiers (e.g. cytokines) within two months of enrollment.
5. Undergone any prostate surgery (e.g. transurethral resection of the prostate (TURP), radical prostatectomy) within two weeks of enrollment.
6. Under the effects of any other hormonal therapy, including anti-androgens for treatment of prostate cancer within three months of baseline.
7. Received leuprolide (leuprorelin) previously.
8. Had an orchiectomy, adrenalectomy or hypophysectomy.
9. Had used any investigational drug, biologic, or device within five half-lives of its physiological action or three months, whichever is longer, before enrollment.
10. Anticipated to need concomitant hormonal, anti-androgen, radiotherapy, chemotherapy, immunotherapy or surgical therapy for prostate cancer throughout the duration of the study.
11. Used over-the-counter (OTC) or alternative medical therapies which has an estrogenic or anti-androgenic effect (e.g., Glycyrrhiza, Dehydroepiandrosterone (DHEA), PC-SPES, saw palmetto) within three months prior to enrollment.
12. Used finasteride, dutasteride, estrogens, megestrol acetate, anti-androgens (Bicalutamide, Flutamide, or Cyproterone), and ketoconazole within three months prior to baseline.
13. Co-existent malignancy or a history of malignancy, with the exception of basal and/or squamous cell carcinomas of the skin.
14. Uncontrolled congestive heart failure within six months before baseline.
15. Experienced a myocardial infarction or a coronary vascular procedure (e.g. balloon angioplasty, coronary artery bypass graft surgery) within six months before baseline.
16. Significant symptomatic cardiovascular disease within six months of baseline.
17. Experienced venous thrombosis within six months of baseline.
18. Uncontrolled hypertension (≥160/100 mmHg) or symptomatic hypotension within three months before baseline.
19. Insulin-dependent diabetes mellitus (Type I diabetes mellitus).
20. History of drug abuse within six months of baseline.
21. Serious intercurrent illnesses or diseases (e.g. hematological, renal, hepatic, respiratory, endocrine, psychiatric) that might interfere with the treatment outlined in the protocol.
22. Receiving anticoagulants or antiplatelet medications and not receiving a stable dose for three months before baseline. Receiving warfarin-derivative anticoagulants with International normalized ratio (INR) outside therapeutic range for the clinical indication for which the anticoagulant has been prescribed.
23. Known hypersensitivity to GnRH, GnRH agonists or any excipients of Leuprolide (leuprorelin).
24. Positive test for HIV, HCV, HbsAg at Screening.
25. History of:

    1. Immunization within four weeks of baseline
    2. Flu shots within two weeks of baseline
    3. Donation or receipt of blood or blood products within two months of baseline
    4. Anaphylaxis
    5. Skin disease which would interfere with injection site evaluation
    6. Dermatographism (Physical urticaria).

Ages: 18 Years to 99 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Testosterone response rate defined as Testosterone values sustained below castration level (0.5 ng/mL or 50 ng/dL) i.e. all Testosterone values at and after Day 28 until Day 57 must be < 0.5 ng/mL or < 50 ng/dL | From Day 28 to day 57

SECONDARY OUTCOMES:
Percentage of subjects who have reached castration level of Testosterone at the last visit (Day 57) | Day 57
Percentage of breakthrough responses defined as a single total serum Testosterone value of >0.5 ng/mL or >50 ng/dL measured after achieving a castration Testosterone level | from Day 28 to Day 57
Time after first implantation until castration level of Testosterone is achieved | up to Day 28
Percentage of subjects with Testosterone values sustained below 0.2 ng/mL or 20 ng/dL at and after Day 28 until Day 57 | From Day 28 to Day 57
Change from baseline in Luteinizing hormone (LH) levels at Day 28 and 57 | from baseline to Day 28 and from baseline to Day 57
Change from baseline in Follicle Stimulating Hormone (FSH) levels at Day 28 and Day 57 | from baseline to Day 28 and from baseline to Day 57
Change from baseline in Prostate-specific antigen (PSA) at Day 57 | Day 57
Mean number of days of maintaining testosterone castration levels (mean number of castration days) | day 28 to day 57
Mean maximum testosterone concentration during the dosing period after reaching the castration level | Day 28 to Day 57

CONTACTS AND LOCATIONS:
Overall Officials: Anirban Roy Chowdhury, Principal Investigator — Bharat Serums and Vaccines Ltd
Locations (2):
- India (2):
  - Government Med ical College & Superspeciality Hospital Nagpur, Nagpur, Maharashtra
  - MV hospital and Research Center, Lucknow, Uttar Pradesh